CLINICAL TRIAL: NCT02523872
Title: Description of Fluid Balance in Patients With Acute Respiratory Failure
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Smiths Medical, ASD, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HP-00064591
Record Dates: First submitted 2015-08-13; First posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Respiratory Insufficiency
Keywords: Fluid overload; Acute respiratory failure; Acute respiratory distress syndrome; Medication administration
MeSH Terms: conditions — Respiratory Insufficiency; Edema; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute respiratory failure: Patients with acute respiratory failure who might benefit from a strategy designed to limit fluid administration

SUMMARY:
The specific aim of this study is to gather data on fluid balance, intravenous medication administration, electrolyte balance, and diuretic and dialysis use in patients with acute respiratory failure who might benefit from a strategy designed to limit fluid administration.

DETAILED DESCRIPTION:
Disruption of fluid balance is common in critical illness. Many critical illnesses are inflammatory in nature and associated with capillary leak and swelling of tissues. While fluid administration may be necessary for the immediate resuscitation of a patient in shock, in the long term it may worsen survival and lead to complications. This is especially true in acute respiratory failure, where excess fluid can lead to a longer duration of mechanical ventilation, longer time in the ICU, and a greater need for dialysis. There is also evidence that conservative fluid administration can prevent complications. Fluid overload is associated with increased healthcare resource utilization and cost.

Much of the fluid administered to patients while in the adult ICU in the United States is administered as medications via large volume infusion pumps. This is a descriptive study to gather data on fluid balance, intravenous medication administration, electrolyte balance, and diuretic and dialysis use in patients with acute respiratory failure who might benefit from a strategy designed to limit fluid administration. The information will be used to design an interventional trial of small volume medication infusion.

ELIGIBILITY:
Inclusion Criteria:

* Intubation and mechanical ventilation for ≤ 7 days
* An underlying condition associated with acute respiratory failure (e.g. pneumonia, ARDS, sepsis, asthma, COPD exacerbation)
* If in shock (MAP < 60, fluid bolus ≥30 ml/Kg or 4 L crystalloid or equivalent, vasopressors except for dopamine ≤ 5 mcg/kg/min or low-dose (≤ 0.04 IU/min) vasopressin) there should be no fluid bolus (1000 mL crystalloid or equivalent) for at least 12 hours

Exclusion Criteria:

* Intubation or mechanical ventilation for > 7 days
* Respiratory failure (requirement for positive pressure ventilation) in past 30 days
* Shock (MAP < 60, fluid bolus ≥30 ml/Kg or 4 L crystalloid or equivalent, vasopressors except for dopamine ≤ 5 mcg/kg/min or low-dose vasopressin) requiring fluid bolus (1000 mL crystalloid or equivalent) within past 12 hours
* Presence of a condition making it unlikely that the patient will be liberated from mechanical ventilation within the next 28 days (e.g. quadriplegia, end-stage lung disease, massive stroke, etc.)
* Prognosis from underlying condition ≤ 28 days (estimated 28 day mortality from underlying condition >50%)
* Likely intention (>50% probability) to withhold or withdraw life-supportive care within next 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute respiratory failure who might benefit from a strategy designed to limit fluid administration
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28 Days
  Discharged from hospital alive or expired
Ventilator-free days | 28 Days
  Number of days of being alive and unassisted breathing by 28 days after time=0
ICU-free days | 28 Days
  Number of days alive and out of ICU-level care by 28 days after time=0
Dialysis use | 28 Days
  Use of intermittent hemodialysis, continuous renal replacement therapy (CvvH, CvvHD), ultrafiltration (intermittent or SCUF), or aquapheresis (Aquadex™)
Sequential Organ Failure Assessment (SOFA) | 28 Days
  Mean and highest scores after T=0

CONTACTS AND LOCATIONS:
Overall Officials: Carl Shanholtz, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Alsous F, Khamiees M, DeGirolamo A, Amoateng-Adjepong Y, Manthous CA. Negative fluid balance predicts survival in patients with septic shock: a retrospective pilot study. Chest. 2000 Jun;117(6):1749-54. doi: 10.1378/chest.117.6.1749. PMID 10858412
- [Background] Maitland K, Kiguli S, Opoka RO, Engoru C, Olupot-Olupot P, Akech SO, Nyeko R, Mtove G, Reyburn H, Lang T, Brent B, Evans JA, Tibenderana JK, Crawley J, Russell EC, Levin M, Babiker AG, Gibb DM; FEAST Trial Group. Mortality after fluid bolus in African children with severe infection. N Engl J Med. 2011 Jun 30;364(26):2483-95. doi: 10.1056/NEJMoa1101549. Epub 2011 May 26. PMID 21615299
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wiedemann HP, Wheeler AP, Bernard GR, Thompson BT, Hayden D, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Comparison of two fluid-management strategies in acute lung injury. N Engl J Med. 2006 Jun 15;354(24):2564-75. doi: 10.1056/NEJMoa062200. Epub 2006 May 21. PMID 16714767
- [Background] Brandstrup B, Tonnesen H, Beier-Holgersen R, Hjortso E, Ording H, Lindorff-Larsen K, Rasmussen MS, Lanng C, Wallin L, Iversen LH, Gramkow CS, Okholm M, Blemmer T, Svendsen PE, Rottensten HH, Thage B, Riis J, Jeppesen IS, Teilum D, Christensen AM, Graungaard B, Pott F; Danish Study Group on Perioperative Fluid Therapy. Effects of intravenous fluid restriction on postoperative complications: comparison of two perioperative fluid regimens: a randomized assessor-blinded multicenter trial. Ann Surg. 2003 Nov;238(5):641-8. doi: 10.1097/01.sla.0000094387.50865.23. PMID 14578723
- [Background] Li G, Malinchoc M, Cartin-Ceba R, Venkata CV, Kor DJ, Peters SG, Hubmayr RD, Gajic O. Eight-year trend of acute respiratory distress syndrome: a population-based study in Olmsted County, Minnesota. Am J Respir Crit Care Med. 2011 Jan 1;183(1):59-66. doi: 10.1164/rccm.201003-0436OC. Epub 2010 Aug 6. PMID 20693377
- [Background] Child DL, Cao Z, Seiberlich LE, Brown H, Greenberg J, Swanson A, Sewall MR, Robinson SB. The costs of fluid overload in the adult intensive care unit: is a small-volume infusion model a proactive solution? Clinicoecon Outcomes Res. 2014 Dec 15;7:1-8. doi: 10.2147/CEOR.S72776. eCollection 2015. PMID 25548524
- [Background] Ferreira FL, Bota DP, Bross A, Melot C, Vincent JL. Serial evaluation of the SOFA score to predict outcome in critically ill patients. JAMA. 2001 Oct 10;286(14):1754-8. doi: 10.1001/jama.286.14.1754. PMID 11594901